CLINICAL TRIAL: NCT05385588
Title: Aging With HIV and Neurocognitive Decline, a Follow-up Study
Acronym: AgingHAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANRS 0093s Aging HAND
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
Keywords: HIV; aging; neurocognitive decline; frailty syndromes
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Prospective study, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): 290 PLHIV, aged 55 to 76 years old
  Interventions: Other: cognitive functional assessment

INTERVENTIONS:
Other: cognitive functional assessment — * Self-administered questionnaire
  * Cognitive and functional tests
  * Medical questionnaire
  * Sampling for biobank (28-32 ml will be collected)

SUMMARY:
The ANRS ( Agence Nationale de Recherches sur le Sida et les Hépatites virales) 0093s Aging HAND study is to assess whether PLHIV (People Living with HIV) initially between 55-70 years of age at baseline analysis under antiretroviral therapy have accelerated decline of neurocognitive function after 6 years of follow-up.

Aging HAND is a French, multicentric, longitudinal, transversal, prospective study with inclusion of 290 PLHIV.

DETAILED DESCRIPTION:
The primary objective of this study is to analyze whether PLHIV initially aged between 55-70 years of age at baseline under antiretroviral therapy have accelerated decline of neurocognitive function after 6 years of follow-up in comparison with an age, gender and educational level matched HIV non-exposed control group from the CONSTANCES cohort.

The secondary objectives of this study are :

* To determine the prevalence of neurocognitive impairment (NCI) according to the Frascati criteria, clinical consensus and alternative classifications, after additional accrual of individuals aged 55 to 76 years for a more precise and extensive age range analysis of NCI
* To describe the incidence and prevalence of the frailty syndromes, and their relation with co-morbidities and NCI, using the Fried score as a measure of frailty
* To constitute a plasma and serum biobank for biomarkers study related to the aging of PLHIV

ELIGIBILITY:
Inclusion criteria

Inclusion criteria for PLHIV for the longitudinal study:

* Having participated in the ANRS EP58 HAND 55-70 study
* A signed informed consent
* To be affiliated and benefit from the French Social Security

Inclusion criteria for PLHIV for the transversal study (only for new subjects):

* HIV-1
* Aged between 55 years and 76 years;
* with a viral load < 50 copies/mL for more than 24 months (with a minimum of 3 available viral loads 6 months prior to inclusion). Blips -defined by a transient increase in viral load- are allowed if < 200 copies/mL, with a maximum of two blips within 24 months;
* With a CD4 (cluster of differentiation 4) count at inclusion ≥ 200 cells/µL for more than the last 12 months (with a last available CD4 count < 6 months of inclusion);
* A signed informed consent
* To be affiliated and benefit from the French Social Security

Exclusion criteria

Non-inclusion criteria for PLHIV for both the longitudinal and transversal studies:

* An Isolated HIV-2 infection
* Confused or with an ongoing neurological disease
* Presenting psychiatric syndromes interfering with cognitive evaluation;
* With sensorial loss, analphabetism or language barriers rendering the interpretation of tests difficult.
* With recent extensive neurocognitive evaluation within 6 months prior to inclusion
* With neurological disease with ongoing clinically relevant sequela
* Participating in another research program, prohibiting the participating in additional research
* Vulnerable: minors, under guardianship or curatorship, or persons deprived of liberty for administrative or judiciary reasons

Ages: 55 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with cognitive decline | 12 months
  The global cognitive decline of patients, expressed through the mean Z-score (with higher scores indicating better cognition) using the mean of z scores of the 5 following cognitive tests (NPZ 5 score): Trail Making Test A-B (TMT A-B), Digit Symbol Substitution Task (DSST) of the WAIS-IV (Wechsler Adult Intelligence Scale), digital finger tapping test, word fluency and formal lexical and semantic evocation for language, Free and Cued Selective Reminding Test.

SECONDARY OUTCOMES:
Proportion of patients with NCI | 12 months
  Presence of neurocognitive impairment (NCI) according to the Frascati criteria and alternative classifications used to define HIV-Associated Neurocognitive Disorder (HAND) in PLHIV
Description of the causes of NCI confirmed | 12 months
  Description of the causes of NCI confirmed after a consensus reached by an expert panel group
Incidence and prevalence of frailty | 12 months
  The Fried frailty score for the ancillary study on incidence and prevalence of frailty

CONTACTS AND LOCATIONS:
Overall Officials: Alain Makinson, Principal Investigator — Department of Infectious and Tropical Diseases, CHU Montpellier
Locations (11):
- France (11):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Saint André, Bordeaux
  - CH Cannes, Cannes
  - CHD Vendée, La Roche-sur-Yon
  - CHU Grenoble Alpes, La Tronche
  - Hôpital Sainte Marguerite, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Carémeau, CHU Nîmes, Nîmes
  - Hopital Pitié Salpêtrière, Paris
  - Hôpital Bretonneau, CHU Tours, Tours